CLINICAL TRIAL: NCT00454363
Title: A Phase 2 Study of GW786034 (Pazopanib) in Advanced Low-Grade or Intermediate-Grade Neuroendocrine Carcinoma
Brief Title: Pazopanib Hydrochloride in Treating Patients With Advanced Neuroendocrine Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00201; NCI-2009-00201 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000537034; MDACC 2006-0077; MDACC 2006-0077 (Other: M D Anderson Cancer Center); 7650 (Other: CTEP); N01CM62202 (NIH); P30CA016672 (NIH); U01CA062490 (NIH)
Record Dates: First submitted 2007-03-27; First posted 2007-03-30 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-03

CONDITIONS: Gastrin-Producing Neuroendocrine Tumor; Lung Carcinoid Tumor; Metastatic Digestive System Neuroendocrine Tumor G1; Multiple Endocrine Neoplasia Type 1; Pancreatic Glucagonoma; Pancreatic Insulinoma; Pancreatic Polypeptide Tumor; Recurrent Digestive System Neuroendocrine Tumor G1; Recurrent Pancreatic Neuroendocrine Carcinoma; Regional Digestive System Neuroendocrine Tumor G1; Somatostatin-Producing Neuroendocrine Tumor
MeSH Terms: conditions — Zollinger-Ellison Syndrome; Multiple Endocrine Neoplasia Type 1; Glucagonoma; Insulinoma; Somatostatinoma | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well pazopanib hydrochloride works in treating patients with advanced neuroendocrine cancer. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the objective response rate (ORR) (complete and partial response) of GW786034 (pazopanib hydrochloride) 800 mg administered orally once daily in patients with advanced low or intermediate grade carcinoid tumors (in carcinoid cohort).

II. To determine the objective response rate (ORR) (complete response and partial response) of GW786034 800mg administered orally once daily in patients with advanced low or intermediate grade pancreatic islet cell carcinoma (in islet cell cohort).

SECONDARY OBJECTIVES:

I. To determine the progression free survival (PFS) duration of GW786034 800mg administered orally once daily in patients with low grade neuroendocrine carcinoma.

II. To determine the safety and tolerability of GW786034 800mg administered orally once daily in patients with low grade neuroendocrine carcinoma.

III. To explore the effect on tumor blood flow as determined by functional computed tomography (CT) of GW786034 800 mg orally once daily in patients with low grade neuroendocrine carcinoma.

IV. To assess the trough level of GW786034 800 mg orally once daily in patients with low grade neuroendocrine carcinoma.

OUTLINE:

Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 90 days for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed low or intermediate grade carcinoid or islet cell carcinoma; patients with carcinoid or islet cell carcinoma associated with multiple endocrine neoplasia (MEN)1 syndrome will be eligible and entered in the islet cell cohort
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Patients may have received 0 or 1 prior cytotoxic therapy; chemotherapy used as a radiosensitizer will be considered one prior chemotherapy regimen; patient must not have received prior bevacizumab or any other therapy targeting vascular endothelial growth factor (VEGF) or VEGF receptors (i.e., SU11248, PTK787/ZK222584, Sorafenib, GW786034)
* Patients must be on a stable dose of somatostatin analogue for 2 months prior to start of protocol; octreotide dose not count toward prior therapy
* Prior radiation therapy is permitted; a recovery period of at least 4 weeks after completion of radiotherapy is required prior to enrollment
* Patients may have received prior interferon (not counted toward prior cytotoxic chemotherapy)
* Patients may have received prior therapy targeting v-kit Hardy-Zuckerman 4 feline sarcoma viral oncogene homolog (c-kit), c-abl oncogene 1, non-receptor tyrosine kinase (abl), platelet-derived growth factor receptor (PDGFR), or epidermal growth factor receptor (EGFR) (imatinib, gefitinib, erlotinib, cetuximab; not counted toward prior cytotoxic chemotherapy)
* Patients must have unresectable or metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, or 1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 120,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 X institutional upper limit of normal
* Creatinine =< 2.0 OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal (calculated by Cockcroft Gault formula)
* Patients must have prothrombin time (PT)/international normalized ratio (INR)/partial thromboplastin time (PTT) within 1.2 X the upper limit of normal
* Patients must have resting blood pressure (BP) no greater than 140 mmHg (systolic) or 90 mmHg (diastolic) for eligibility; initiation or adjustment of BP medication is permitted prior to study entry
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation; women of child-bearing potential must have a negative blood pregnancy test prior to study entry; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:

  * An intrauterine device with a documented failure rate of less than 1% per year
  * Vasectomized partner who is sterile prior to the female patient's entry and is the sole sexual partner for that female
  * Complete abstinence from sexual intercourse for 14 days before exposure to investigation product, through the clinical trial, and for at least 21 days after the last dose of investigational product
  * Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide)

    * Note: Oral contraceptives are not reliable due to potential drug-drug interaction
* Ability to understand and the willingness to sign a written informed consent document
* Ability to swallow and retain oral medication

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks prior to study enrollment; at least 4 weeks must have elapsed since any major surgery prior to study enrollment
* Patients may not be receiving any other investigational agents
* Patients with corrected QT (QTc) > 480 msecs
* Patients with greater than 1+ (>= 100 mg/dl) proteinuria on two consecutive routine urinalysis taken at least 1 week apart are ineligible
* Certain medications that act through the cytochrome P450 (CYP450) system are specifically prohibited in patients receiving GW786034 (pazopanib) because in vitro data indicate that the agent has the potential to interact with the cytochrome P450 isoenzymes; certain other agents should be used with caution
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for intravenous [IV] alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain GW786034 (pazopanib) tablets are excluded
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
  * History of known active diverticulitis within the past 3 months
  * Any history of cerebrovascular accident (CVA) within the last 6 months
  * Current use of therapeutic warfarin; Note: Low molecular weight heparin and prophylactic low-dose warfarin are permitted; PT/PTT must meet the inclusion criteria
  * History of myocardial infarction, cardiac arrhythmia, admission for unstable angina, cardiac angioplasty or stenting within the last 12 weeks
  * History of venous thrombosis in last 12 weeks
  * Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system; a patient who has a history of class II heart failure and is asymptomatic on treatment may be considered eligible
* Patients with known brain metastases should be excluded from this clinical trial
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, or any other cancer from which the patient has been disease free for five years
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with GW786034 (pazopanib); these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Uncontrolled diarrhea (8 or more bowel movements per day)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-03; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Yao, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Phan AT, Halperin DM, Chan JA, Fogelman DR, Hess KR, Malinowski P, Regan E, Ng CS, Yao JC, Kulke MH. Pazopanib and depot octreotide in advanced, well-differentiated neuroendocrine tumours: a multicentre, single-group, phase 2 study. Lancet Oncol. 2015 Jun;16(6):695-703. doi: 10.1016/S1470-2045(15)70136-1. Epub 2015 May 5. PMID 25956795

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open recruitment period: March 2007 to December 2009. All recruitment done at University of Texas (UT) and Dana Farber Cancer Institute.
Pre-assignment Details: Of the 52 enrolled, one participant was excluded from the study prior to study treatment.
Groups:
- Pazopanib + Carcinoid: Carcinoid Tumor Type: Oral Pazopanib hydrochloride 800 mg once daily on days 1-28.
- Pazopanib + pNET: Pancreatic Neuroendocrine (pNET) tumor type: Oral Pazopanib hydrochloride 800 mg once daily on days 1-28.
Period: Overall Study
Arm/Group | Pazopanib + Carcinoid | Pazopanib + pNET
Started | 20 | 31
Completed | 15 | 29
Not Completed | 5 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal prior to 12 weeks treatment | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pazopanib + Carcinoid | Pazopanib + pNET | Total
Number analyzed (Participants) | 20 | 31 | 51
Age, Continuous [Median (Full Range); unit: years] | 63 [43 to 79] | 55 [34 to 77] | 60 [34 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 13 | 21 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 18 | 28 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 20 | 28 | 48
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 31 | 51
Participant from Enrolling Institutions [Number; unit: participants]
  Dana Farber Cancer Institute | 6 | 11 | 17
  MD Anderson Cancer Center | 14 | 20 | 34

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (Complete and Partial Response) for Each Cohort Assessed by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: RECIST Criteria: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): 30% decrease in sum of longest diameter (LD) of target lesions, reference baseline sum LD; Progressive Disease (PD): 20% increase in sum of LD of target lesions, reference smallest sum LD recorded since treatment started or appearance 1/> new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum LD since treatment started.
Time Frame: Up to 18 months
Population: RECIST best protocol response by intention to treat. Four participants were not evaluable for response.
Measure: Number; unit: participants
Arm/Group | Pazopanib + Carcinoid | Pazopanib + pNET
Number analyzed (Participants) | 20 | 31
participants
  PR | 0 | 6
  SD | 14 | 21
  PD | 3 | 3
  Not Evaluable | 3 | 1

2. Secondary Outcome: Percent Change in Tumor Blood Flow Assessed by Functional CT
Description: Explore the effect on tumor blood flow as determined by functional CT of GW786034 (Pazopanib) 800 mg orally once daily on both arms, carcinoid and pNET.
Time Frame: Baseline and week 12
Population: Data were not collected from any participant in the Pazopanib + Carcinoid Arm Group
Measure: Median (Full Range); unit: percentage of change in tumor blood flow
Arm/Group | Pazopanib + Carcinoid | Pazopanib + pNET
Number analyzed (Participants) | 0 | 11
percentage of change in tumor blood flow |  | 139 [-56 to 154]

3. Other Pre Specified Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death.
Time Frame: Baseline to 18 months.
Population: Analysis calculated according to intent to treat.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib + Carcinoid | Pazopanib + pNET
Number analyzed (Participants) | 20 | 31
months | 12 [3.4 to 20.6] | 14.2 [6.9 to 21.5]

4. Other Pre Specified Outcome: Plasma Trough Level of GW786034
Time Frame: assessed at Baseline and day 28, day 28 reported
Population: Plasma trough level in blood was below the level of detection.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib + Carcinoid | Pazopanib + pNET
Number analyzed (Participants) | 20 | 31
Participants | NA — Plasma trough level in blood was below the level of detection. | NA — Plasma trough level in blood was below the level of detection.

ADVERSE EVENTS:
Time Frame: Adverse events occurring within 30 days of last dose investigational drug, with each cycle 28 days for up to 12 cycles. Overall participation period April 2007 to March 2013.
Groups:
- Pazopanib: Oral pazopanib hydrochloride once daily on days 1-28.
Arm/Group | Pazopanib
Serious Adverse Events (participants affected / at risk) | 16/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib (N=51)
Death NOS (General disorders) | 11
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Thromboembolic event (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pazopanib (N=51)
Abdominal distension (Gastrointestinal disorders) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 36 (78)
Acidosis (Metabolism and nutrition disorders) | 2 (4)
Activated partial thromboplastin time prolonged (Blood and lymphatic system disorders) | 5 (10)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 19 (58)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 9 (28)
Allergic rhinitis (Immune system disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 23 (45)
Anorexia (Gastrointestinal disorders) | 12 (14)
Anxiety (Nervous system disorders) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7)
Ascites (Gastrointestinal disorders) | 3 (3)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 27 (83)
Back Pain (Musculoskeletal and connective tissue disorders) | 12 (15)
Bladder Spasm (Renal and urinary disorders) | 1 (1)
Blood bilirubin increased (Metabolism and nutrition disorders) | 17 (33)
Blurred vision (Eye disorders) | 3 (3)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cardiac disorders (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Cholesterol high (Metabolism and nutrition disorders) | 3 (3)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Nervous system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 15 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Creatinine increased (Metabolism and nutrition disorders) | 5 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Depression (Nervous system disorders) | 5 (6)
Diarrhea (Gastrointestinal disorders) | 41 (150)
Dizziness (Nervous system disorders) | 11 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Edema, Face (General disorders) | 1 (1)
Edema, Limbs (General disorders) | 8 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 1 (1)
Eye infection/pain (Eye disorders) | 2 (2)
Fatigue (General disorders) | 43 (155)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 10 (13)
Flatulence (Gastrointestinal disorders) | 3 (3)
Flushing (Skin and subcutaneous tissue disorders) | 7 (11)
Gastritis (Gastrointestinal disorders) | 14 (17)
Administration site issue (Injury, poisoning and procedural complications) | 1 (2)
Headache (Nervous system disorders) | 14 (26)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 3 (6)
Hot flashes (Endocrine disorders) | 3 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 23 (73)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 3 (5)
Hypertension (Cardiac disorders) | 35 (45)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 6 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (15)
Hypoglycemia (Metabolism and nutrition disorders) | 4 (11)
Hypokalemia (Metabolism and nutrition disorders) | 4 (8)
Hypomagnesemia (Metabolism and nutrition disorders) | 10 (15)
Hyponatremia (Metabolism and nutrition disorders) | 6 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (9)
Hypotension (Cardiac disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 3 (3)
Infections (Infections and infestations) | 5 (5)
INR increased (Blood and lymphatic system disorders) | 8 (16) — International Normalized Ratio (INR) of prothrombin time
Insomnia (General disorders) | 11 (12)
Investigations (Investigations) | 2 (3)
Libido decreased (Reproductive system and breast disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 10 (21)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle Weakness, Trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (General disorders) | 3 (4)
Nail Loss (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 37 (104)
Nervous system disorders (Nervous system disorders) | 3 (3)
Neuralgia (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 11 (29)
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Oral pain (Gastrointestinal disorders) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 20 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (7)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 3 (5)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 12 (19)
Proteinuria (Metabolism and nutrition disorders) | 7 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 (6)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin disorders (Skin and subcutaneous tissue disorders) | 8 (10)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 7 (7)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (2)
Syncope (Nervous system disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Increased Urinary Frequency (Renal and urinary disorders) | 6 (7)
Urinary Incontinence (Renal and urinary disorders) | 1 (1)
Urine Retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vaginal infection (Reproductive system and breast disorders) | 2 (2)
Vasovagal reaction (Cardiac disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (2)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Vomiting (Gastrointestinal disorders) | 20 (37)
Weight gain (General disorders) | 2 (2)
Weight loss (General disorders) | 8 (10)
White blood cell decreased (Blood and lymphatic system disorders) | 10 (19)
Wound dehiscence (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less